CLINICAL TRIAL: NCT01901861
Title: Effect of a Single Dose of the DPP-4 Inhibitor on Islet Function After Igestion of a Standardized Mixed Meal in Subjects With Type 2 Diabetes
Brief Title: Effect of the DPP-4 Inhibitor Sitagliptin on Islet Function After Mixed Meal in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Bo Ahren, professor, Lund University
Allocation: Non-Randomized | Model: Factorial | Masking: None
Other Study IDs: 2012-005660-98
Record Dates: First submitted 2013-07-14; First posted 2013-07-17 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes
Keywords: GLP-1, GIP, DPP-4 inhibition, iset function
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sitagliptin (Active Comparator): Sitagliptin 100mg is given before meal ingestion
  Interventions: Drug: Sitagliptin
- Placebo (Placebo Comparator): Placebo is given before meal ingestion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100mg is given before meal ingestion
  Other Names: Mixed meal test with sitagliptin
  Arms: Sitagliptin
Drug: Placebo — Placebo is given before meal ingestion
  Other Names: Mixed meal test with placebo
  Arms: Placebo

SUMMARY:
study hypothesis to examine the acute effects on glycaemia and islet hormone secretion of increased levels of endogenous GLP-1 and GIP on islet cell function in men with type 2 diabetes. To this purpose, a standardized mixed meal test will be ingested with or without concomitant administration of sitagliptin (100mg).

DETAILED DESCRIPTION:
In men subjects with type 2 diabetes treated with diet and exercise with or without metformin treatment as an antidiabetic agent, a standardized mixed meal test will be served with or without administration of sitagliptin (100mg).

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men with type 2 diabetes diagnosed according to ICD10
* Ongoing treatment with life style adjustment or life style adjustment together with metformin as oral antidiabetic. Metformin therapy should not exceed 2 grams daily
* Age 20-75 years
* HbA1c ≤80 mmol/mol
* BMI: 20-40 kg/m2

Exclusion Criteria:

* Liver disease or ALAT three times above upper reference range
* Diabetic nephropathy (GFR < 50 mL/min/1.73 m2 or albuminuria)
* Proliferative diabetic retinopathy
* Treatment with any glucose-lowering medication except metformin
* Previous myocardial infarction, coronary heart disease or insatiable angina pectoris in the last 6 months.
* Previous surgery on the gastrointestinal tract
* Larger surgical intervention during the last 12 weeks
* Treatment with oral steroids or thiazide diuretics
* Treatment with digoxin
* Smokers
* Participation in another study the last 4 weeks
* Paracetamol intolerance

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Release of incretins hormones | 300 min

CONTACTS AND LOCATIONS:
Overall Officials: Bo Ahren, Professor, Principal Investigator — Lund University
Locations (1):
- Department of Clinical Science Lund,Lund University, Lund, Sweden